CLINICAL TRIAL: NCT05902741
Title: The Impact of a Race-Based Stress Reduction Intervention on Well-Being, Inflammation, and DNA Methylation in African American Women at Risk for Cardiometabolic Disease
Brief Title: The Impact of a Race-Based Stress Reduction Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Karen Saban, Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 214133
Record Dates: First submitted 2023-05-02; First posted 2023-06-15 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-07

CONDITIONS: Racism; Stress; Inflammation
MeSH Terms: conditions — Racism; Inflammation

STUDY DESIGN:
Intervention Model Description: Self-identified African American women will be randomized to either the race-based stress reduction intervention group (Resilience, Stress, and Ethnicity [RiSE]) or the HEP.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resilience, Stress, and Ethnicity (RiSE) program (Experimental): Resilience, Stress, and Ethnicity (RiSE) program is an 8-session weekly group-based intervention that integrates cognitive-behavioral strategies focused on the biopsychosocial impact of racism, racial identity development, and empowerment. RiSE has three primary components:
  1. processing and sharing experiences related to race based stress,
  2. psychoeducation on the biopsychosocial impact of racism,
  3. skill building and empowerment.
  Interventions: Behavioral: RiSE
- Health Education Program (HEP) (Active Comparator): Health Education Program
  Interventions: Behavioral: HEP

INTERVENTIONS:
Behavioral: RiSE — RiSE provides participants with a platform to share the emotional impact of race-based stress and to offer supportive listening to their peers. Participants explicitly discuss the experiences they have as African American women, taking into account the ways which the interaction between their racial and gender identities shapes their experiences. Facilitators review difficulties associated with addressing racism and unique experiences of Black women at interpersonal and structural levels, and provide evidence of strategies to promote effective communication and internal emotional regulation regarding experiences of racism. Facilitators provide psychoeducation on intersectionality, structural racism, overt racism, microaggressions, and internalized racism. Following this education, facilitators help participants utilize cognitive-behavioral strategies to understand consequent thoughts, feelings, and actions associated with such experiences.
  Arms: Resilience, Stress, and Ethnicity (RiSE) program
Behavioral: HEP — The HEP group will consist of classes focusing on wellness promotion. Expert speakers provide the HEP classes (e.g dietician, pharmacist).
  Arms: Health Education Program (HEP)

SUMMARY:
The goal of this clinical trial is to learn whether a stress reduction program called Resilience, Stress, and Ethnicity (RiSE) improves well-being, inflammation, and the epigenome in African American (AA) women who have risk factors for heart or metabolic disease.

The main question it aims to answer is whether an intervention that integrates cognitive-behavioral strategies focused on the impact that social stress, such as racism, has on the body, racial identity development, and empowerment.

Participants will placed in one of the two following groups:

* The RiSE program will focus on teaching participants how to reduce their stress levels and will meet online weekly for approximately 2 hours each week for 8 consecutive weeks.
* The Health Education program will include education on how to improve general health and will meet online weekly for approximately 2 hours each week for 8 consecutive weeks.

Participants will provide saliva to measure cytokines and DNA methylation (DNAm), complete questionnaires, and have blood pressure, heart rate, and weight measured at the following clinic visits:

1. Prior to starting the intervention
2. Mid-way through the intervention (Week 4)
3. End of the intervention (Week 8)
4. Six (6) months after the completion of the intervention

DETAILED DESCRIPTION:
Participants of both programs - RiSE and Health Education Program (HEP) - will meet weekly for 8 consecutive weeks for approximately 2 hours every week. Two booster sessions will occur one month and two months after completion of the interventions. Classes will meet synchronously over Zoom. RiSE classes will be facilitated by two trained clinical psychologists. Expert speakers will be hired to provide the HEP classes (e.g dietician, pharmacist). The investigators will vary the time of day for each 8- week program in order to meet the scheduling needs of participants. Cohorts of 9-12 participants each and sessions for the treatment and control group will be provided concurrently. Topics for the health education program (HEP) (attention-control) were selected so they would not confound the overall objectives of the RiSE program.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 50 and 75
* Female
* Post-menopausal (without menstrual period for at least 12 consecutive months)
* Self-identified AA or Black
* Able to write, read, speak English
* Must have at least 1 of any of the following:

  * Waist circumference >88 cm
  * Systolic BP>130 mmHg and/ or diastolic BP>88 mmHg or on antihypertensive medications
  * Diagnosed and/or being treated for hypercholesterolemia
  * History of Type 2 diabetes

Exclusion Criteria:

* History of myocardial infarction or ischemic heart disease/angina, stent placement, coronary artery bypass, left ventricular hypertrophy, congestive heart failure, or ischemic stroke
* Any major immune-related disease (e.g., rheumatoid arthritis. lupus)
* Use of immune-altering medications, such as glucocorticoids
* Periodontal disease, bleeding gums, dental work in past 72 hours
* Current smoker or has smoked in past 3 months
* Active cancer
* Active infection
* Substance abuse
* Cognitive or psychiatric disorder that would affect ability to participate in classes (Brief Screen for Cognitive Impairment total score of 8 or higher)

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified African American women
Enrollment: 300 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Current perceived stress | 8 months
  Perceived Stress Scale (PSS-10). Scores range from 0 to 40 with higher score suggesting worse outcome.

SECONDARY OUTCOMES:
General coping | 8 months
  Ways of Coping Questionnaire. Scores range for 0 to 198 for total scale with higher scores suggesting more coping.
Coping with discrimination | 8 months
  Coping with Discrimination Scale. Scores range from 25 to 150 with higher scores suggesting more coping.
Internalized racism | 8 months
  Appropriated Racial Oppression Scale. Scores range from 24 to 168 with higher score suggesting worse outcome.
Resistance and empowerment | 8 months
  Resistance and Empowerment Against Racism Scale. Scores range from 26 to 130 with higher score suggesting better outcome.
DNA methylation | 8 months
  Targeted DNA methylation of targeted candidate genes
Stress overload | 8 months
  Stress Overload Scale. Scores range from 30 to 150 with higher score suggesting worse outcome.
Depressive symptoms | 8 months
  Beck Depression Inventory (BDI). Scores range from 0 to 63 with higher score suggesting worse outcome.
Anxiety | 8 months
  Generalized Anxiety Disorder-7 (GAD-7). Scores range from 0 to 21 with higher score suggesting worse outcome.
Fatigue | 8 months
  NIH Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form 8a
Sleep disturbance | 8 months
  NIH PROMIS Short Form v1.0
Inflammatory burden- C-reactive protein (CRP) | 8 months
  Salivary CRP
Inflammatory burden - Tumor necrosis factor-alpha (TNF-alpha) | 8 months
  Salivary TNF-alpha
Inflammatory burden - Interleukin-6 (IL-6) | 8 months
  Salivary IL-6
Inflammatory burden - Interleukin-1 beta (IL-1B) | 8 months
  Salivary IL-1B
Inflammatory burden - Interferon gamma (IFN-γ), | 8 months
  Salivary IFN-y

CONTACTS AND LOCATIONS:
Overall Officials: Karen Saban, RN, PhD, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University Chicago, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Genomic data will be individual level data. Analysis of genomic DNA will link genotype to phenotypic information obtained as part of this study. Genomic data will include Genome wide association (GWAS) and DNA methylation (EWAS). Genomic data will be obtained from saliva taken at baseline, at completion of intervention, and 6 months after completion of intervention.
  The protocol, sample informed consent, case report forms, data dictionary, and code book will be made accessible in data repositories where data are shared. For data submitted to Database of Genotypes and Phenotypes (dbGaP), variable-level metadata will be provided using details of Common Data Elements, definitions, and standards used for data collection and sharing.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: The repository will make the data accessible within 3 years of last participant study visit or at the end of the performance period, or no later than the date of online publication, whichever is soon.
  Genomic data will be shared according to Genomic Data Sharing (GDS) policy, which requires that genomic data must be submitted within 3 months following data generation, and released within 6 months of data submission to the repository or at acceptance of the publication, whichever is first. Data will be preserved within the repository for at least three years following the completion of the grant, as required by federal retention guidelines.
Access Criteria: Data will be shared with controlled access in the dbGAP for non-commercial research use by qualified investigators, as allowed by the participants' informed consent and the Institutional Certification. Due to ethical considerations, access to the resulting scientific data will be limited and approved by the Multiple Principal Investigators (MPI) Saban and Taylor.

REFERENCES:
- [Derived] Saban KL, Joyce C, Nyembwe A, Janusek L, Tell D, de la Pena P, Motley D, Shawahin L, Prescott L, Potts-Thompson S, Taylor JY. The Effectiveness of a Race-Based Stress Reduction Intervention on Improving Stress-Related Symptoms and Inflammation in African American Women at Risk for Cardiometabolic Disease: Protocol for Recruitment and Intervention for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Apr 18;14:e65649. doi: 10.2196/65649. PMID 40250840